CLINICAL TRIAL: NCT03613376
Title: Compression And Functional Ability After Endovenous Varicose Vein Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Toni Pihlaja, Vascular specialist, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 97/2018
Record Dates: First submitted 2018-05-27; First posted 2018-08-03 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Varicose Veins of Lower Limb; Varicose Veins
Keywords: Varicose veins; Compression stockings; Sclerotherapy; Radiofrequency ablation
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Compression (No Intervention): Patients in this group will not receive any compression after treatment
- Compression (Active Comparator): Patients in this group will use class II compression stockings continuously until next evening and then next 4 days during daytime.
  Interventions: Other: Class II compression stockings

INTERVENTIONS:
Other: Class II compression stockings — Patients in this group will use class II compression stocking continuously until next evening and then next 4 days during daytime
  Arms: Compression

SUMMARY:
Study's aim is to study possible differences in post-operative rehabilitation, functional ability and visual disturbances after endovascular varicose intervention (RF-catheter and foam sclerotherapy) in two study groups, where patients will be randomised to either no compression group (Group I) or compression group (Group II)

ELIGIBILITY:
Inclusion Criteria:

* Duplex ultrasound verified GSV, AASV and/or SSV incompetence suitable for radiofrequency ablation
* Comprehensive Classification System for Chronic Venous Disorders (CEAP) rated from C2 to C4
* Distal varicose vein insufficiency suitable for sclerotherapy
* Patient willingness to participate

Exclusion Criteria:

* History of pulmonary embolism or deep venous thrombosis
* Large (>12mm) truncal vein diameter
* CEAP C5-C6
* Antithrombotic medication (ASA accepted)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 10days recorded daily
  Visual Analog Scale (VAS) 0-100mm

SECONDARY OUTCOMES:
Functional ability, other than pain | 10 days recorded daily
  Visual Analog Scale 0-100mm indicating post-operative functional ability reduction
Aberdeen Varicose Veins Questionnaire (AVVQ) | Assessed preoperatively and at 2 months
  Score from 0 to 99.658
Visual appearance of varicose veins, patient assessment | Preoperatively and at 2 months
  Patient self-assessment (Patient Self-Assessment of Visible Varicose Veins, PA-V score)
Signs of deep venous thrombosis hematoma | Assessed at 2 months and earlier if necessary
  Ultrasound assessment
Time required returning to normal activity | 14 days
Time required returning to full activity | 14 days
Postoperative pigmentation | at 2 months
  Pigmentation is monitored from standardised photographs on severity of pigmentation and most severe tone of post-operative pigmentation compared to base skin colour, reviewers are blinded to study group.
Visual appearance of varicose veins, expert assessment | Preoperatively and at 2 months
  Photography Review -Visible Varicose Veins (IPR-V score, reviewers are blinded to time point and study group).

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Vascular Department, Oulu, Finland